CLINICAL TRIAL: NCT06114654
Title: Gluteal Musculature Activation to Improve Ankle Stability: a Cross-sectional Observational Study
Brief Title: Gluteal Musculature Activation to Improve Ankle Stability
Acronym: TOBEMG
Status: Completed | Type: Observational
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, CRISTINA ADILLÓN, Principal Investigator, University Rovira i Virgili
Other Study IDs: 074/2022
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Ankle Disease; Muscle Weakness
Keywords: biomechanics; electromyography; ankle stability; gluteal musculature
MeSH Terms: conditions — Muscle Weakness | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Physiotherapy students of the Rovira i Virgili University aged between 18 and 35 years enrolled during the academic year 2022-2023. All participants were allowed three practice trials for each test. Consistent feedback was provided throughout to ensure proper technique. Electrodes were placed to assess muscle activity according to SENIAM recommendations in gluteus medius, gluteus maximus, tibialis anterior and peroneus longus. After electrode placement, a maximal isometric strength test (MVIC) was performed for each muscle to normalize the electromyographic data. During this MVIC test, the maximum isometric force was measured using the Chronojump Boscosystem force gauge. Following this, ankle stability evaluation tests were performed. The Single Leg Stance Test, the Hurdle Step test and finally the Single leg vertical jump will be performed.
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Physical Therapy — Specific physical tests to assess muscle strength, ankle stability and activation of the lower extremity musculature: Single Leg Stance Test, Hurdle Step test and Single leg vertical jump.

SUMMARY:
The goal of this observational study is to to evaluate and correlate muscle activation in the gluteal musculature and ankle stability in a healthy population. The main question it aims to answer is: Is there a significant positive correlation between gluteal muscle activation and ankle stability?

Participants will complete questionnaires on the functionality of foot and ankle pathologies related to their daily life and sports activities, and perform specific physical tests to assess muscle strength, ankle stability, and activation of the lower extremity musculature.

DETAILED DESCRIPTION:
The main outcomes were the muscle activation (gluteus maximus, gluteus medius, tibialis anterior, and peroneus longus) of both limbs during a Single Leg Stance test and a Hurdle Step test (Check Your Motion, Albacete, Spain). Muscle activation was assessed using surface electromyography, and the results will be described as a percentage of Maximum Isometric Voluntary Contraction (%MVIC). Ankle stability was evaluated according to the criteria established by Perrot using a force platform (Dynamic Walkway P6000, BTS Bioengineering, Milan, Italy).

There are no previous studies evaluating a possible correlation between gluteus maximus muscle activity and ankle stabilization capacity. Therefore, a sample size calculation was performed with the aim of detecting a strong correlation as statistically significant (r=0.5) according to the criteria of Hopkins et al [33]. The G*Power 3.1 program was used to calculate the sample size. The statistical test used was "Correlation: Bivariate Normal Model", the type of power analysis was "A priori: compute required sample size - given alpha, power and effect size". An error α=0.05 and a statistical power of 0.80 (β=0.20) was used. The result of the test was 29 subjects required to perform this research.

The study investigators will sign a data confidentiality sheet where they commit to use the data with appropriate confidentiality. In addition, after analyzing the results, the participant's face will be hidden so that he/she cannot be recognized.

The data will be collected on a form designed for this purpose and will be entered into a database created with the Microsoft Office Excel® 2021 program, in a URV system subject to the security measures of the National Security Scheme, always in areas where only the research staff of this project can access. Subsequently, the SPSS program (Statistical Package for the Social Sciences) version 26.0 for Windows® will be used to analyze the data.

The normality of all variables will be examined using the Saphiro Wilk statistical test. Descriptive statistics for all variables will be expressed as mean (standard deviation) if the variable follows a normal distribution and as median (interquartile range) if the variable does not follow a normal distribution. Subsequently, correlation analysis will be performed using Pearson's correlation test (if both variables are normal) or Spearman's Rho (if either variable does not follow a normal distribution). Correlations will be classified as weak (r=0.1), moderate (r=0.3), strong (r=0.5), large (r=0.7) or very large (r=0.9) [33]. Correlations will be described as statistically significant if the p-value is less than 0.05. If the correlation coefficient is statistically significant, the coefficient of determination (R2) will be calculated. Bonferroni correction for multiple comparisons will be applied based on the correlations finally evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18 and 35 years of age.
* To sign the informed consent form.
* Failure to meet the exclusion criteria.

Exclusion Criteria:

* To have an injury at the time of selection.
* To have psychological and/or psychiatric illnesses.
* To take anticoagulants, to have an infectious process.
* To have a heart disease.
* To be hypersensitive to pain.
* To have skin infections.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health students from the Faculty of Medicine and Health Sciences of the Rovira i Virgili University.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Muscle activation (%MVIC) | 1 year
  This was measured with wireless electromyography sensors electromiografía (BTS FreeEMG 1000, BTS Bioengineering, Milan, Italy).
Ankle stability | 1 year
  This was measured with force platform (Dynamic Walkway P6000, BTS Bioengineering, Milan, Italy).

SECONDARY OUTCOMES:
Aye | 1 year
  Years
Gender | 1 year
  Female or male
Height | 1 year
  Centimeters
Body weight | 1 year
  Kilograms
Ankle functionality | 1 year
  This was measured with a Foot and Ankle Ability Measures questionnaire. It consists of 9 items, each item has a certain score and the sum of these should give a result between 0 and 30 points. If the result is ≤ 27 points, it indicates ankle instability.
Maximum isometric muscle strength | 1 year
  This was measured with a force gauge, Chronojump Boscosystem

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Adillón, PhD, Principal Investigator — University Rovira i Virgili
Locations (1):
- Rovira i Virgili University, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No